CLINICAL TRIAL: NCT06987123
Title: Toripalimab in Combination With Capecitabine as Adjuvant Therapy After Surgery for Locally Recurrent Resectable Nasopharyngeal Carcinoma: a Single-arm Clinical Trial
Brief Title: TC as Adjuvant Therapy After Surgery for Locally Recurrent Resectable Nasopharyngeal Carcinoma: a Single-arm Clinical Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, YiJun Hua, Chief Physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-FXY-459-NPC
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
Keywords: recurrent nasopharyngeal carcinoma; salvage surgery; Toripalimab; capecitabine
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — toripalimab; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Toripalimab in combination with capecitabine as adjuvant therapy after surgery for locally recurrent resectable nasopharyngeal carcinoma
  Interventions: Drug: Toripalimab; Drug: Capecitabine; Procedure: salvage surgery

INTERVENTIONS:
Drug: Toripalimab — Toripalimab 240 mg, administered on the first day, Q3W × 17 cycles
Drug: Capecitabine — Capecitabine 650 mg/m2 twice a day, oral administration, d1-21, Q3W × 17 cycles
Procedure: salvage surgery — The specific steps of high-frequency electrosurgical knife treatment for localized recurrent nasopharyngeal carcinoma are as follows:
  1. It must be performed under general anesthesia, with the complete resection of the nasopharyngeal tumor and its sufficient safe boundary through both nasal cavities under the guidance of nasal endoscopy. When marking the surgical margin, the anterior margin should reach 1-2cm in front of the posterior column of the nasal septum, and the upper margin can reach about 0.5-1cm to the upper margin of the posterior nostril. The lateral and lower margins are designed individually based on the size and location of the tumor. The basic principle is to ensure a safe margin of 0.5-1.0cm, and then use low-temperature plasma ablation. Ablate the tumor tissue and the normal tissue at the resection margin layer by layer from the upper resection margin to the lower resection margin until no obvious tumor residue was observed with the naked eye.
  2. Rinse the surgical c

SUMMARY:
Regarding the application value of capecitabine metronome chemotherapy's regulatory effect on the immune microenvironment in nasopharyngeal carcinoma, many studies in recent years have confirmed that metronome chemotherapy and immunotherapy are safe and effective in resectable recurrent nasopharyngeal carcinoma. Therefore, the investigators plan to conduct a "single-arm clinical study on adjuvant therapy of toripalimab combined with capecitabine after Surgery for locally recurrent resectable nasopharyngeal carcinoma" to explore the efficacy and safety of toripalimab combined with capecitabine as adjuvant therapy after salvage surgery for resectable recurrent nasopharyngeal carcinoma. If this study is confirmed, it is expected to provide a new treatment model for patients with resectable recurrent nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Regarding the application value of capecitabine metronome chemotherapy's regulatory effect on the immune microenvironment in nasopharyngeal carcinoma, many studies in recent years have confirmed that metronome chemotherapy and immunotherapy are safe and effective in resectable recurrent nasopharyngeal carcinoma. Therefore, the investigators plan to conduct a "single-arm clinical study on adjuvant therapy of toripalimab combined with capecitabine after Surgery for locally recurrent resectable nasopharyngeal carcinoma" to explore the efficacy and safety of toripalimab combined with capecitabine as adjuvant therapy after salvage surgery for resectable recurrent nasopharyngeal carcinoma. If this study is confirmed, it is expected to provide a new treatment model for patients with resectable recurrent nasopharyngeal carcinoma.The diagnosis was pathologically confirmed as locally recurrent nasopharyngeal carcinoma. According to the TNM staging of recurrent nasopharyngeal carcinoma (AJCC, 8th Edition, 2018), resectable nasopharyngeal diseases: rT1 (the tumor was confined to the nasopharynx, oropharynx and/or nasal cavity, and did not involve the parapharynx); rT2 (The tumor is confined to the superficial septum beside the pharynx, more than 0.5 cm away from the internal carotid artery) and rT3 (the tumor is confined to the basal wall of the sphenoid sinus, more than 0.5 cm away from the internal carotid artery and the cavernous sinus); Resectable recurrent regional lymph nodes (rN1-3), without involvement of the anterior vertebral fascia, cervical vertebrae or common carotid artery/internal carotid artery.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed as locally recurrent nasopharyngeal carcinoma, according to the TNM staging of recurrent nasopharyngeal carcinoma (AJCC, 8th Edition, 2018), resectable nasopharyngeal diseases: rT1 (the tumor is confined to the nasopharynx, oropharynx and/or nasal cavity, and does not involve the parapharynx); rT2 (The tumor is confined to the superficial septum beside the pharynx, more than 0.5 cm away from the internal carotid artery) and rT3 (the tumor is confined to the basal wall of the sphenoid sinus, more than 0.5 cm away from the internal carotid artery and the cavernous sinus); Resectable recurrent regional lymph nodes (rN1-3), without involvement of the anterior vertebral fascia, cervical vertebrae or common carotid artery/internal carotid artery.
* It has been more than 6 months since the last radiotherapy
* Age: 18-70 years old, gender not limited;
* ECOG score: 0-1 point;
* The functions of the major organs are normal, that is, the following standards are met; (1) The blood routine examination standards must meet (no blood transfusion or blood products within 14 days) : a. HB≥90 g/L; b. ANC≥1.5×109/L; c. PLT≥80×109/L; (2) Biochemical tests must meet the following standards: a. TBIL<1.5× upper normal limit (ULN); b. ALT and AST<2.5×ULN; c. Serum Cr≤1.5×ULN or endogenous creatinine clearance rate > 45 ml/min;
* Women of childbearing age should agree to use contraceptive measures during the study period and within 6 months after the end of the study (e.g Intrauterine devices, contraceptive pills or condoms; The serum or urine pregnancy test must be negative within 7 days before enrollment in the study, and the patient must be a non-lactating patient. Male patients who should agree that contraceptive measures must be adopted during the study period and within 6 months after the end of the study period;
* Sign the informed consent form and voluntarily participate in the clinical trial research project.

Exclusion Criteria:

* The tumor broke through the dura mater at the base of the skull and severely involved the brain parenchyma, with distant metastasis and obvious complications, and the patient could not be under general anesthesia.
* Patients with tumor recurrence or residual after re-radiotherapy.
* The patient has any active autoimmune diseases or a history of autoimmune diseases (such as the following, but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism; Vitiligo Asthma that requires medical intervention with bronchodilators;
* Patients who are currently undergoing immunosuppressive therapy with immunosuppressants or systemic hormones to achieve the purpose of immunosuppression (dose >10mg/ day prednisone or other therapeutic hormones) and are still continuing to use them within 2 weeks before enrollment;
* Have received immunotherapy within the past six months;
* Patients with any severe and/or uncontrollable diseases, including: those with unsatisfactory blood pressure control (systolic) Patients with blood pressure >=160mmHg or diastolic blood pressure >=100 mmHg; Suffering from grade II or above myocardial ischemia or myocardial infarction, arrhythmia (including QT interval >=480ms), and grade II cardiac insufficiency; Active or uncontrolled severe infection; Liver diseases such as decompensated liver disease, active hepatitis B (HBV-DNA>=104 copy number /ml or 2000IU/ml) or hepatitis C (positive hepatitis C antibody and HCV-RNA higher than the detection limit of the analytical method);
* Pregnant or lactating women; Patients with other malignant tumors within 8.5 years (except for cured basal cell carcinoma of the skin and cervical carcinoma in situ);
* Those with a history of abuse of psychotropic drugs and who are unable to quit or those with mental disorders;
* Patients who have participated in clinical trials of other similar drugs within three months;
* According to the researcher's judgment, there are concomitant diseases that seriously endanger the patient's safety or affect the patient's completion of the study;
* Those that the researchers consider unsuitable for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-05-18 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  2-year progression-free survival

IPD SHARING:
Plan to Share IPD: No
Researchers who has been approveed can share.